CLINICAL TRIAL: NCT05540288
Title: NAlmefene Versus Placebo in Addition to Treatment as Usual on Craving in Behavioural Addictions
Acronym: NABAb
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC21_0336
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Behavioural Addiction
Keywords: Nalmefene; Craving; Behavioural addiction; Gambling disorder; Food addiction; Sexual addiction
MeSH Terms: conditions — Gambling; Food Addiction; Compulsive Sexual Behavior Disorder | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nalmefene (Experimental)
  Interventions: Drug: Nalmefene
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nalmefene — Week 1: 18 mg/d
  Week 2:
  1. In the absence of ARs or in the presence of grade 1 or 2 ARs, 36 mg/d
  2. In the presence of grade 3 ARs, 18 mg/d
  3. In the presence of grade 4 ARs, treatment will be stopped immediately.
  Week 3 to week 5:
  1. In case of acceptable safety profile at the 18mg/d dosage during week 2, the treatment will be maintained at the same dosage
  2. In the presence of sustained grade 3 ARs at the 18mg/d dosage during week 2, the treatment will be stopped.
  3. In case of acceptable safety profile at the 36mg/d dosage during week 2, the treatment will be maintained at the same dosage
  4. In the presence of grade 3 ARs at the 36mg/d dosage during week 2, the treatment dosage will be decreased at 18mg/d
  5. Whatever the dosage during week 2, in the presence of grade 4 ARs, the treatment will be stopped immediately.
  Arms: Nalmefene
Drug: Placebo — Week 1: 1 tablet/d
  Week 2:
  1. In the absence of ARs or in the presence of grade 1 or 2 ARs, 2 tablets/d
  2. In the presence of grade 3 ARs, 1 tablet/d
  3. In the presence of grade 4 ARs, the treatment will be stopped immediately.
  Week 3 to week 5:
  1. In case of acceptable safety profile at the dosage of 1 tablet/d during week 2, the treatment will be maintained at the same dosage
  2. In the presence of sustained grade 3 ARs at the dosage of 1 tablet/d during week 2, the treatment will be stopped.
  3. In case of acceptable safety profile at the dosage of 2 tablets/d during week 2, the treatment will be maintained at the same dosage
  4. In the presence of grade 3 ARs at the dosage of 2 tablets/d during week 2, the treatment dosage will be decreased at 1 tablet/d
  5. Whatever the dosage during week 2, in the presence of grade 4 ARs, the treatment will be stopped immediately.
  Arms: Placebo

SUMMARY:
Behavioural addictions (BAs) [gambling disorder (GD), food addiction (FA), sexual addiction (SA)] may lead to disastrous consequences. They are often associated with other addictive or psychiatric disorders, and high rates of suicide attempts. Epidemiological studies report prevalence reaching 2.7% for GD, 5% for SA, and up to 7.9% for FA.

Many similarities have been highlighted between BAs, as well as with substance use disorders. One core clinical similarity between those disorders is craving (uncontrollable urge to engage in rewarding behaviours), which has been consistently associated with diminished control over the behaviour and relapse.

At present, no pharmacological treatment has been approved for BAs, but several medications have been tested. Among them, two opioid receptor antagonists - naltrexone and nalmefene - appear the most promising. By decreasing dopamine neurotransmission in the reward circuitry, they reduce both excitement for rewarding behaviours and craving.

Compared to naltrexone, nalmefene seems to have a better safety. To date, no study investigated the efficacy of nalmefene as a pan-addiction treatment for BAs. Two clinical trials have demonstrated its efficacy for the treatment of GD, but no clinical trial was conducted for FA and SA.

The investigators hypothesise that nalmefene (36 mg/d), compared to a placebo, can have a therapeutic effect as an add-on to usual treatment for decreasing craving in several BAs.

ELIGIBILITY:
Pre-inclusion Criteria:

* Males and females ≥ 18 years old
* Patient already in care or newly initiating care in Addictology departments for a beharioural addiction, diagnosed with current:

  * Gambling disorder [NORC DSM Screen for Gambling Problems (NODS), revised for DSM-5]
  * Food addiction [Yale Food Addiction Scale (YFAS), revised for DSM-5]
  * Or Sexual addiction [interview adapted from the NODS to explore the diagnostic criteria proposed by Carnes et al. (2012): NODS-SA]
* Able to regularly assess and report their craving episodes on a weekly diary
* Who provide their written informed consent
* Affiliated with French social security system or beneficiary from such system

Inclusion Criteria:

* Having presented at least one episode of craving with an intensity ≥ 4/10 at the NRS during the week prior to inclusion

Women must meet one of the following criteria at the time of inclusion:

* use adequate contraceptive measures as recommended by the CTFG (Recommendations related to contraception and pregnancy testing in clinical trials v1.1), and have a negative pregnancy test (urine test) prior to receiving the first dose of study drug;
* or be post-menopausal (over 50 years of age with amenorrhea for at least 12 months after discontinuation of all exogenous hormonal therapy)
* or (if under 50 years of age) have been amenorrheic for at least 12 months after discontinuation of exogenous hormonal therapy and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels corresponding to post-menopausal levels
* or have undergone irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy (this operation must be documented).

Exclusion Criteria:

* Being currently treated by another anti-craving drug that have been already tested for craving reduction in BAs (naltrexone, acamprosate, baclofène, topiramate, bupropion, N-acetyl-cystéine, disulfiram, etc.);
* Presenting a contraindication for the use of nalmefene (listed in the SmPC):

  * Known hypersensitivity to the active substance or to any of the excipients. In particular, intolerance to galactose or deficiency in Lapp lactase or glucose-galactose malabsorption (rare hereditary diseases);
  * Treatment by opioid agonists (full or partial) (opioid pain relievers, opioid substitution drugs);
  * Recent history of opioid dependence or current opioid dependence;
  * Current symptoms of the acute opioid withdrawal syndrome;
  * Suspected recent consumption of opioid (necessity to consider the half-life);
  * Severe hepatic impairment (Child-Pugh stage B or C);
  * Severe renal impairment (estimated glomerular filtration rate [TFGe] <30 mL/min/1.73 m2);
  * History of recent acute alcohol withdrawal syndrome (including hallucinations, convulsions and delirium tremens).
* Predictable opioid treatment during the study period;
* Unstable psychiatric disorders (meaning disorders for which the treatment was modified since less than a month (corresponding to the instauration of a new treatment, or the increase in dosage of a treatment already being taken)), including severe risk of suicide (i.e. necessity to engage specific medication or hospitalization; psychotropic medication engaged since less than 1 month; absence of improvement after one month of medication) (because nalmefene has not been studied in patients with unstable psychiatric disorders). Patients with a food addiction diagnosed with eating disorders marked by the presence of binge eating can be included;
* Anorexia nervosa-restricting type (because food addiction concept is poorly established among patients with AN-R, who do not have binge eating episodes induced by craving);
* Extreme leanness (body mass index < 16.5) (because loss of appetite and/or weight loss are frequent adverse effects of nalmefene);
* Current treatment with potent inhibitor drugs of the UGT2B7 (UDP-Glucuronosyltransferase-2B7); for example: diclofenac, fluconazole, medroxyprogesterone acetate, meclofenamic acid;
* Current treatment with UGT inducing drugs; for example: dexamethasone, phenobarbital, rifampicin, omeprazole;
* Inability to indicate the time of day of the most intense craving episode (because this information will determine the time of day the treatment should be taken);
* Pregnancy (attested by a pregnancy urinary test for women of childbearing age) or breastfeeding woman;
* Trusteeship;
* Major cognitive impairment;
* Not fluent in French;
* Participation to another interventional study during the last month or expected participation to another interventional study during participation to the NABAB study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Variation of averaged intensity of craving episodes between start and end of treatment. | 5 weeks
  Variation of averaged intensity of craving episodes between start (during the week preceding initiation of treatment) and end (during the week preceding end of treatment) of treatment. Each craving episode will be reported by the patient on a weekly diary, with intensity assessed through a Numerical Rating Scale (NRS) form 0 to 10 (0=lowest intensity and 10= highest intensity).

SECONDARY OUTCOMES:
Variation of averaged weekly frequency (number of episodes) of craving episodes between start and end of treatment. | 5 weeks
Variation of averaged weekly duration (cumulative duration of all episodes) of craving episodes between start and end of treatment. | 5 weeks
Variation of averaged weekly intensity, frequency and duration of craving episodes between start of treatment and 4 weeks after the end of treatment. | 9 weeks (5 weeks of treatment +4 weeks of follow up after treatment)
Variation of averaged weekly frequency of the BA episodes: (i) between start and end of treatment and (ii) between start of treatment and 4 weeks after the end of treatment. | 9 weeks
Variation of averaged weekly duration of the BA episodes: (i) between start and end of treatment and (ii) between start of treatment and 4 weeks after the end of treatment. | 9 weeks
Variation of averaged weekly intensity of the BA episodes: (i) between start and end of treatment and (ii) between start of treatment and 4 weeks after the end of treatment. | 9 weeks
  Assessed through a Numerical Rating Scale (NRS) form 0 (lowest intensity) to 10 (highest intensity)
Overall clinical improvement, assessed though the Clinical Global Impression - Improvement (CGI-I) scale. | 9 weeks
Overall clinical improvement, assessed though the GGI - Efficacy Index (CGI-EI). | 9 weeks
Variation of averaged weekly use of psychoactive substances (including nicotine) and daily life behaviors of interest (gambling, sex, food) between start of treatment and 4 weeks after the end of treatment | 9 weeks
Number, type and severity of self-reported adverse side effects, during either weeks of treatment at a dosage of 18 mg/d or 36 mg/d. | 9 weeks
Mutation(s) associated with non-response to nalmefene treatment | 9 weeks
Sociodemographic, medical and clinical data, especially psychiatric and addictive co-morbidities assessed with the Mini International Neuropsychiatric Interview - Simplified (MINI-S) and the age of the BA | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL-BRONNEC, Principal Investigator — Nantes University Hospital
Locations (13):
- France (13):
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CH de La Rochelle, La Rochelle
  - Hospices Civils de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHRU de Tours, Tours
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided